CLINICAL TRIAL: NCT04272632
Title: Coload Optimization Guided by Inferior Vena Cava Collapsibility Index in Parturients With Prophylactic Norepinephrine Infusion Undergoing Cesarean Section: a Randomized, Dose-finding Trial
Brief Title: Coload Optimization Guided by Inferior Vena Cava Collapsibility Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2020-3
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-02

CONDITIONS: Adverse Effect
Keywords: Coload; Inferior vena cava collapsibility index; Norepinephrine; Cesarean section; Dose-finding
MeSH Terms: interventions — Population Groups; Crystalloid Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4 ml/kg group (Experimental): 4 ml/kg compound sodium chloride (0.85% NaCl, 0.03% KCl, and 0.033% CaCl2) was given immediately after spinal anesthesia.
  Interventions: Drug: 4 ml/kg group
- 8 ml/kg group (Experimental): 8 ml/kg compound sodium chloride (0.85% NaCl, 0.03% KCl, and 0.033% CaCl2) was given immediately after spinal anesthesia.
  Interventions: Drug: 8 ml/kg group
- 12 ml/kg group (Experimental): 12 ml/kg compound sodium chloride (0.85% NaCl, 0.03% KCl, and 0.033% CaCl2) was given immediately after spinal anesthesia.
  Interventions: Drug: 12 ml/kg group

INTERVENTIONS:
Drug: 4 ml/kg group — 4 ml/kg compound sodium chloride (0.85% NaCl, 0.03% KCl, and 0.033% CaCl2) was given immediately after spinal anesthesia.
  Other Names: Crystalloid
  Arms: 4 ml/kg group
Drug: 8 ml/kg group — 8 ml/kg compound sodium chloride (0.85% NaCl, 0.03% KCl, and 0.033% CaCl2) was given immediately after spinal anesthesia.
  Other Names: Crystalloid
  Arms: 8 ml/kg group
Drug: 12 ml/kg group — 12 ml/kg compound sodium chloride (0.85% NaCl, 0.03% KCl, and 0.033% CaCl2) was given immediately after spinal anesthesia.
  Other Names: Crystalloid
  Arms: 12 ml/kg group

SUMMARY:
The purpose of this study is to investigate the optimal coload guided by inferior vena cava collapsibility index in parturients with prophylactic norepinephrine infusion undergoing cesarean section.

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. Vasopressors has been highly recommended for routine prevention and/or treatment of post-spinal anesthesia hypotension. As a potential substitute drug for phenylephrine, norepinephrine has gradually been used in parturients undergoing cesarean section. There's some evidence that prophylactic infusion of norepinephrine could effectively reduce the incidence of post-spinal anesthesia hypotension in parturients undergoing cesarean section. However, our study (NCT03997500) had been shown that inferior vena cava collapsibility index (IVC-CI) markedly decreased in prophylactic norepinephrine infusion versus normal saline after spinal anesthesia and fetal delivery, suggesting that more prudent fluid management is required. The ideal dose of coload and coload is still unknown. Thus, the purpose of this study is to investigate the optimal coload guided by IVC-CI in parturients with prophylactic norepinephrine infusion undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years
* Primipara or multipara
* Singleton pregnancy ≥37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for elective cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥ 160mmHg
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
The minimum (IVC-min), maximum diameter (IVC-max) and collapsibility index (IVC-CI) of the inferior vena cava (IVC) | Baseline (before preload)
  IVC-CI = [(IVC-max-IVC-min) /IVC-max*100%]
The minimum (IVC-min), maximum diameter (IVC-max) and collapsibility index (IVC-CI) of the inferior vena cava (IVC) | Before spinal anesthesia (after preload)
  IVC-CI = [(IVC-max-IVC-min) /IVC-max*100%]
The minimum (IVC-min), maximum diameter (IVC-max) and collapsibility index (IVC-CI) of the inferior vena cava (IVC) | 5 min after spinal anesthesia
  IVC-CI = [(IVC-max-IVC-min) /IVC-max*100%]
The minimum (IVC-min), maximum diameter (IVC-max) and collapsibility index (IVC-CI) of the inferior vena cava (IVC) | 5 min after fetal delivery
  IVC-CI = [(IVC-max-IVC-min) /IVC-max*100%]
The minimum (IVC-min), maximum diameter (IVC-max) and collapsibility index (IVC-CI) of the inferior vena cava (IVC) | Before leaving the operating room
  IVC-CI = [(IVC-max-IVC-min) /IVC-max*100%]

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline.
The incidence of severe post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of bradycardia | 1-15 minutes after spinal anesthesia
  Heart rate < 55 beats/min.
The incidence of hypertension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline
pH | Immediately after delivery
  From umbilical vein blood gases
Partial pressure of oxygen | Immediately after delivery
  From umbilical vein blood gases
Base excess | Immediately after delivery
  From umbilical vein blood gases
APGAR score | 1min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
Overall stability of systolic blood pressure control versus baseline | 1-15 minutes after spinal anesthesia.
  Evaluated by performance error (PE).
Overall stability of heart rate control versus baseline | 1-15 minutes after spinal anesthesia.
  Evaluated by performance error (PE).

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Ni, Dr., Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China